CLINICAL TRIAL: NCT02883842
Title: Effectiveness of Text Messaging on Risk Factors Control and Medication Adherence Among Patients With Coronary Heart Disease and Diabetes in China: Cardiovascular Health and Text Messaging-Diabetes Mellitus (CHAT-DM) Study
Brief Title: Cardiovascular Health and Text Messaging-Diabetes Mellitus (CHAT-DM) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201502009-2
Record Dates: First submitted 2016-08-24; First posted 2016-08-30 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease; Diabetes
Keywords: Coronary artery disease; Diabetes; Text messages
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention-Text messaging (Experimental): Patients will receive regular semi-personalized text messages for 6 months. Each participants will receive 6 text messages per week, which will be sent at random times of the day (9.00am, 12noon, 4.00pm). They will receive one general messages, one hypertension message, one glucose control message, one lifestyle message, one medication adherence message and one physical activity message per week.
  Interventions: Behavioral: Text messaging
- Control (No Intervention): Participants in the control group will receive 2 thank-you messages per month and undertake routine clinical practice.

INTERVENTIONS:
Behavioral: Text messaging — Patients will receive regular semi-personalized text messages for 6 months. Each participants will receive 6 text messages per week, which will be sent at random times of the day (9.00am, 12noon, 4.00pm). They will receive one general messages, one hypertension message, one glucose control message, one lifestyle message, one medication adherence message and one physical activity message per week. Prior to study commencement, a bank of 270 messages have been developed based on guidelines and behavior change theory (BCT), and have underwent multidisciplinary expert review and qualitative review process.
  Arms: Intervention-Text messaging

SUMMARY:
The study is a two-arm, parallel, randomized clinical trial. The purpose of the study is to evaluate the effectiveness of automated mobile phone text message-based intervention for secondary prevention, including lifestyles modification, medication adherence improvement and risk factors control among coronary heart disease (CHD) patients with diabetes. The participants will be randomized into intervention and control groups in a 1:1 ratio. The intervention group will receive 6 pre-designed text messages per week in addition to usual care for 6 months, while the control group will receive usual care.

DETAILED DESCRIPTION:
Objective: This study aims to evaluate the effectiveness of automated mobile phone text message-based intervention for secondary prevention, including lifestyles modification, medication adherence improvement and risk factors control among CHD patients with diabetes. We hypothesized that an intervention using mobile phone text based education and reminder can improve risk factors control and medication adherence for CHD patients.

Study design: The study is a two-arm, parallel, randomized clinical trial. Patients will be eligible if they have documented CHD defined as having history of myocardial infarction and percutaneous coronary intervention (PCI), have a history of diabetes mellitus, have the capability of reading and sending short message, and are able to provide informed consent. Patients will be excluded if they do not have an active mobile phone. The eligible participants will be allocated into intervention and control groups in a 1:1 ratio randomly. The intervention group will receive intervention of pre-designed text messages in addition to usual care, while the control group will receive usual care. All the participants will be followed up for 6 months.

Study intervention: Participants in the intervention group will receive text messages for 6 months as well as usual care. They will receive one general messages, one hypertension message, one glucose control message, one lifestyle message, one medication adherence message and one physical activity message per week.

Outcome measures: The primary endpoint is the change in glycemic hemoglobin (HbA1C) as measured by central blood sample. Secondary endpoints include a change in proportion of patients achieving HbA1C<7%, body mass index (BMI), physical activity, medication adherence, systolic blood pressure, low-density lipoprotein cholesterol (LDL-C) and fasting blood glucose (FBG). Exploratory endpoints include long-term prognosis of the patients, such as death, nonfatal myocardial infarction, stroke and so on, as well as health status (SAQ and EQ-5D).

Statistical analysis: Evaluation will be carried out on an intention-to-treat basis. Values of analyzed endpoints between intervention group and control group will be compared according to the analysis plan. We'll follow a prespecified analysis plan and subgroup analysis will be conducted accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Participants with coronary artery disease defined as history of myocardial infarction and PCI
* History of diabetes
* Capability to read and send text messages

Exclusion Criteria:

* Assumed poor adherence
* Do not have an active mobile phone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in glucose level measured by HbA1C level | Baseline; 6 months
  We will measured the change in glucose level from baseline to 6 months.

SECONDARY OUTCOMES:
Change in proportion of patients achieving HbA1C<7% | Baseline; 6 months
  We will measure the change in proportion of patients achieving HbA1C<7% from baseline to 6 months.
Change in level of fasting blood glucose (FBG) | Baseline; 6 months
  We will measure the change in FBG level from baseline to 6 months.
Change in body mass index (BMI) according to national standards | Baseline; 6 months
  We will measured the change in BMI from baseline to 6 months.
Change in systolic blood pressure (SBP) obtained in office during each interview | Baseline; 6 months
  We will measured the change in SBP from baseline to 6 months.
Change in level of physical activity measured via International Physical Activity Questionnaire (IPAQ) scale | Baseline; 6 months
  We will measure the change in IPAQ scale from baseline to 6 months.
Change in medication adherence | Baseline; 6 months
  We will measure the change in medication adherence from baseline to 6 months.
Change in low-density lipoprotein cholesterol (LDL-C) level | Baseline; 6 months
  We will measure the change in LDL-C level from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, MD, PhD, Principal Investigator — China National Center for Cardiovascular Disease; Harlan M Krumholz, MD, SM, Principal Investigator — Yale University
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huo X, Krumholz HM, Bai X, Spatz ES, Ding Q, Horak P, Zhao W, Gong Q, Zhang H, Yan X, Sun Y, Liu J, Wu X, Guan W, Wang X, Li J, Li X, Spertus JA, Masoudi FA, Zheng X. Effects of Mobile Text Messaging on Glycemic Control in Patients With Coronary Heart Disease and Diabetes Mellitus: A Randomized Clinical Trial. Circ Cardiovasc Qual Outcomes. 2019 Sep;12(9):e005805. doi: 10.1161/CIRCOUTCOMES.119.005805. Epub 2019 Aug 31. PMID 31474119
- [Derived] Huo X, Spatz ES, Ding Q, Horak P, Zheng X, Masters C, Zhang H, Irwin ML, Yan X, Guan W, Li J, Li X, Spertus JA, Masoudi FA, Krumholz HM, Jiang L. Design and rationale of the Cardiovascular Health and Text Messaging (CHAT) Study and the CHAT-Diabetes Mellitus (CHAT-DM) Study: two randomised controlled trials of text messaging to improve secondary prevention for coronary heart disease and diabetes. BMJ Open. 2017 Dec 21;7(12):e018302. doi: 10.1136/bmjopen-2017-018302. PMID 29273661